CLINICAL TRIAL: NCT06435936
Title: A Phase 1 Double-Blinded, Randomized, Placebo-Controlled Study Assessing Safety and Pharmacokinetics of Intramuscular SAB-176 (a Tc Bovine Derived Anti-Influenza Human Immunoglobulin) in Healthy Subjects
Brief Title: A Study to Assess the Safety of SAB-176 to Prevent the Flu, Given IM in Healthy Adults Compared With Placebo
Acronym: SAB-176-103
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SAb Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: SAB-176-103
Record Dates: First submitted 2024-05-14; First posted 2024-05-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: PHA1A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- SAB-176 1 mL (Experimental): 1 mL (~75 mg) SAB-176 dose
  Interventions: Drug: Single Ascending Dose of SAB-176
- Placebo 1mL (Placebo Comparator): Normal Saline
  Interventions: Drug: Single Ascending Dose of Placebo
- SAB-176 3mL (Experimental): 3 mL (~225 mg) SAB-176 dose
  Interventions: Drug: Single Ascending Dose of SAB-176
- Placebo 3mL (Placebo Comparator): Normal Saline
  Interventions: Drug: Single Ascending Dose of Placebo
- SAB-176 5mL (Experimental): 5 mL (~375 mg) SAB-176 dose
  Interventions: Drug: Single Ascending Dose of SAB-176
- Placebo 5mL (Placebo Comparator): Normal Saline
  Interventions: Drug: Single Ascending Dose of Placebo
- SAB-176 20mL (Experimental): 20 mL (~1500 mg) SAB-176 dose
  Interventions: Drug: Single Ascending Dose of SAB-176
- Placebo 20mL (Placebo Comparator): Normal Saline
  Interventions: Drug: Single Ascending Dose of Placebo

INTERVENTIONS:
Drug: Single Ascending Dose of SAB-176 — Single ascending dose
  Other Names: SAB-176
  Arms: SAB-176 1 mL; SAB-176 20mL; SAB-176 3mL; SAB-176 5mL
Drug: Single Ascending Dose of Placebo — Single ascending dose
  Other Names: Placebo
  Arms: Placebo 1mL; Placebo 20mL; Placebo 3mL; Placebo 5mL

SUMMARY:
This study will evaluate the safety and tolerability of an intramuscular injection of SAB-176 intended for use as a pre/post prophylactic for influenza.

This is a Phase 1, randomized, double-blind, placebo-controlled clinical trial in which a total of 28 subjects will receive an injection of either SAB-176 or placebo (normal saline). The investigational product will be administered intramuscularly (IM) on Day 1. Four dose escalation cohorts of 7 subjects (5 active and 2 placebo) each are planned. Subjects will be randomized to receive either SAB-176 or placebo in a double-blinded manner.

Progression to subsequent dose-escalating cohorts will be dependent on safety measured through Day 5 after dosing of the previous cohort.

Blood specimens will be collected at prescribed intervals to examine pharmacokinetics and immunogenicity. Safety will be actively monitored during investigational product administration and for 60 days following dosing. The decision to advance to the next cohort will be based solely on the safety assessment through Day 5. All safety data will be summarized and reviewed by the PI, the Sponsor's Clinical Monitor, and the Research Monitor prior to next cohort dose-escalation.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety of an experimental product for influenza. Influenza, commonly known as the flu, causes substantial illness and death worldwide despite available treatments and vaccines. The U.S. military is susceptible to large outbreaks from new strains of influenza and effective treatment options can be limited. Importantly, the DoD deploys people all over the world. Flu treatment may be more limited overseas. Thus, the military is trying to develop new products to treat and prevent influenza.

The experimental product being testing in this study is called SAB-176. It was developed by SAB Biotherapeutics, Inc. SAB-176 is an immunoglobulin product designed to prevent the flu and/or reduce its symptoms. Immunoglobulins are antibodies (disease fighting substances) made by the immune system that can prevent and treat infections. SAB-176 comes from the plasma (the light yellow liquid part of blood) of immunized cows. Antibodies in the plasma are collected and purified. Those purified antibodies are SAB-176.

This study will assess the safety of the experimental study product, SAB-176, in healthy adults. SAB-176 is not approved by the U.S. Food and Drug Administration (FDA) yet and is investigational. The FDA is aware of this trial though and this research is required before SAB- 176 can be approved. SAB-176 will be given by intramuscular injection (a shot into the muscle). The study is designed to find out if it is safe to give increasing doses of SAB-176. The investigators will look for any side effects. The study will also assess the amount of SAB-176 circulating in participant's bloodstream. The investigators want to find a safe dose of SAB-176 that also enables SAB-176 to circulate in the blood for a longer time. The investigators think this will provide longer lasting protection against the flu. Some participants will be given a placebo instead of SAB-176. The placebo contains normal saline (salt water). The placebo does not contain any of the active ingredients of SAB-176. The investigator and sponsor will compare the side effects of those who got the placebo to those who got SAB-176. This helps to know which side effects are caused by SAB-176. Neither Participants nor the study staff will know what Participants are getting until after the study is complete. Participants will be assigned to receive either SAB-176 or the placebo randomly (like rolling dice).

Participants will be in the study for about 3 months. Participants will need to attend a screening visit to determine if Participants are eligible to participate. If Participants are eligible and Participants agree to join the study, Participants will remain in the study for 2 months after Participants receive SAB-176 or placebo to monitor any side effects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy adult, male or female, aged 18 to 60 years (inclusive) at the time of enrollment.

  2. Completion and review of assessment of understanding test (achieved > 70% accuracy).

  3. Signed informed consent document. 4. Available for the required follow-up period and scheduled clinic visits. 5. Women of childbearing potential: Negative urine pregnancy test with understanding (through informed consent process) to not become pregnant during the study or within two (2) months following investigational product administration.

  6. Willing to use an acceptable method of contraception during the study and for 2 months following investigational product administration. If a barrier method is the contraceptive of choice, concurrent use of a spermicide will be recommended.

  7. Body mass index (BMI) between 19 and 35 kg/m2. 8. Agree to refrain from blood donation during the study and for at least 12 months (1 year) following injection with the study drug.

Exclusion Criteria:

* 1. Health problems (for example, intercurrent febrile illness, chronic medical conditions such as psychiatric conditions, diabetes mellitus, hypertension, or any other condition that might place the subject at increased risk of adverse events); study clinicians, in consultation with the PI, will use clinical judgment on a case-by-case basis to assess safety risks under this criterion.

  2. Clinically significant abnormalities on physical examination that, in the PI's opinion, would place the subject at undue risk and/or preclude full evaluation of potential adverse events.

  3. Immunosuppressive drugs (use of systemic corticosteroids or chemotherapeutics that may influence antibody development) or inherited or acquired immunodeficiency (including IgA deficiency; defined by serum IgA <7 mg/dL).

  4. Women who are pregnant or planning to become pregnant during the study period plus 2 months beyond the last received dose, and currently nursing women.

  5. History of buttock enhancement (e.g., silicone enhancement or implants) that may interfere with intramuscular injections.

  6. Participation in research involving another investigational product (defined as receipt of an investigational product such as a drug or vaccine or exposure to an invasive investigational device) within 30 days prior to dosing or any time through the last study safety visit.

  7. Receipt of any unapproved immunizations or vaccines within 30 days prior to planned dosing.

  8. Positive blood test for HBsAg, HCV, or HIV-1/2. 9. Clinically significant abnormalities on basic laboratory screening. 10. Moderate or severe influenza requiring hospitalization in the 30 days prior to planned dosing.

  11. Receipt of any blood product (e.g., RhoGam, IVIG) within 120 days prior to planned dosing.

  12. Use of other drugs that, in the opinion of the investigator, could complicate the safety assessment of SAB-176 (e.g., medications or over-the-counter vitamins or supplements formulated in bovine gelatin).

  13. Vaccination against influenza less than 90 days prior to product administration.

  14. Known autoimmune condition requiring therapy more intensive than intermittent nonsteroidal anti-inflammatories in the 6 months prior to planned dosing (e.g., rheumatoid arthritis, lupus, inflammatory bowel disease).

  15. Chronic respiratory disease including chronic obstructive pulmonary disease (COPD), emphysema, cystic fibrosis, pulmonary hypertension, or other chronic condition that requires the routine use of supplemental oxygen.

  16. Chronic asthma requiring the use of oral steroids or hospitalization in the last six months; inhaled steroids are permitted.

  17. Receipt of pooled immunoglobulin or plasma within 30 days prior to planned dosing.

  18. History of allergy, anaphylaxis, or severe reaction to beef products (including dairy products and gelatin).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of solicited local and systemic adverse events (AEs) through Day 29. | Dosing through Day 29
  Solicited AEs will be collected after administration of the investigational product up to 28 days post-injection. Unsolicited AEs will be collected until the last study visit (up to Day 61). AEs will be summarized for the number of subjects who experience an AE or the number of AE events by analysis group, MedDRA category, severity grading scale, and post-baseline timepoint.
Occurrence of IP-related unsolicited AEs through Day 61. | Dosing through Day 61
  Solicited AEs will be collected after administration of the investigational product up to 28 days post-injection. Unsolicited AEs will be collected until the last study visit (up to Day 61). AEs will be summarized for the number of subjects who experience an AE or the number of AE events by analysis group, MedDRA category, severity grading scale, and post-baseline timepoint.
Occurrence of serious adverse events (SAEs) through Day 61. | Dosing through Day 61
  Solicited AEs will be collected after administration of the investigational product up to 28 days post-injection. Unsolicited AEs will be collected until the last study visit (up to Day 61). AEs will be summarized for the number of subjects who experience an AE or the number of AE events by analysis group, MedDRA category, severity grading scale, and post-baseline timepoint.

SECONDARY OUTCOMES:
Hemagglutination Inhibition (HAI) against influenza A strains (H1N1, H3N2) | 1 hour post dose, Day 1, Day 8, Day 14, Day 28, Day 60
  The pharmacokinetic profile will be assessed based on hemagglutination inhibition against multiple influenza A strains (H1N1, H3N2).
Microneutralization (MN) titers against influenza A strains (H1N1, H3N2) | 1 hour post dose, Day 1, Day 8, Day 14, Day 28, Day 60
  The pharmacokinetic profile will be assessed based on microneutralization against multiple influenza A strains (H1N1, H3N2).
Hemagglutination Inhibition (HAI) against influenza B strains (B-Victoria lineage, B/Yamagata lineage) | 1 hour post dose, Day 1, Day 8, Day 14, Day 28, Day 60
  The pharmacokinetic profile will be assessed based on hemagglutination inhibition against influenza B strains (B-Victoria lineage, B/Yamagata lineage).
Microneutralization (MN) titers against influenza B strains (B-Victoria lineage, B/Yamagata lineage) | 1 hour post dose, Day 1, Day 8, Day 14, Day 28, Day 60
  The pharmacokinetic profile will be assessed based on microneutralization against influenza B strains (B-Victoria lineage, B/Yamagata lineage).
Maximum titer value (Cmax) | 1 hour post dose, Day 1, Day 8, Day 14, Day 28, Day 60
  The pharmacokinetic profile will be assessed using the following parameter: maximum titer value (Cmax)
Time of maximum titer value (Tmax) | 1 hour post dose, Day 1, Day 8, Day 14, Day 28, Day 60
  The pharmacokinetic profile will be assessed using the following parameter: time of maximum titer value (Tmax)
Terminal phase elimination rate constant (λZ) | 1 hour post dose, Day 1, Day 8, Day 14, Day 28, Day 60
  The pharmacokinetic profile will be assessed using the following parameter: terminal phase elimination rate constant (λZ)
Terminal elimination half-life (t½) | 1 hour post dose, Day 1, Day 8, Day 14, Day 28, Day 60
  The pharmacokinetic profile will be assessed using the following parameter: terminal elimination half-life (t½).
Area under the curve (AUC) | 1 hour post dose, Day 1, Day 8, Day 14, Day 28, Day 60
  The pharmacokinetic profile will be assessed using the following parameter: area under the curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Nehkonti Adams, MD, Principal Investigator — Naval Medical Research Command (NMRC)
Locations (1):
- Naval Medical Research Command (NMRC), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No